CLINICAL TRIAL: NCT00005994
Title: Patient Information and Antiemetic Drug Efficacy
Brief Title: Patient Education in Preventing Nausea and Vomiting in Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Gary Morrow, Director, URCC CCOP Research Base, University of Rochester
Allocation: Randomized
Other Study IDs: CDR0000067996; URCC-3996; NCI-P00-0160
Record Dates: First submitted 2000-07-05; First posted 2004-06-09 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Nausea and Vomiting; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: nausea and vomiting; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ondansetron

INTERVENTIONS:
Drug: ondansetron

SUMMARY:
RATIONALE: Patient education may improve the effectiveness of ondansetron in preventing nausea and vomiting in patients receiving chemotherapy.

PURPOSE: This randomized clinical trial is studying how well patient education works in preventing nausea and vomiting in cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether an educational intervention to enhance the effectiveness of ondansetron can prevent acute postchemotherapy nausea and emesis in cancer patients. II. Assess any potential effectiveness of the intervention on delayed postchemotherapy nausea and emesis in these patients. III. Examine the effect of the intervention on patient expectations.

OUTLINE: This is a randomized, double blind, multicenter study. Patients are stratified by center and chemotherapy agent (cisplatin vs carboplatin vs doxorubicin). Patients are randomized to one of two treatment arms. Arm I: Patients receive standard educational materials. Arm II: Patients receive specific intervention material in addition to standard educational materials. Patients then complete a patient information questionnaire. Patients receive ondansetron orally or IV over 10-15 minutes in addition to the first 2 courses of chemotherapy. Patients complete a nausea and emesis questionnaire after each of their first 2 chemotherapy treatments.

PROJECTED ACCRUAL: A total of 300 patients (150 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Chemotherapy naive with diagnosis of any cancer scheduled to receive chemotherapy containing cisplatin, carboplatin, or doxorubicin

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary R. Morrow, PhD, MS, Study Chair — James P. Wilmot Cancer Center
Locations (4):
- United States (4):
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Rochester Cancer Center, Rochester, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina